CLINICAL TRIAL: NCT04492423
Title: VerifyNow® PRUTest® Cardiovascular Population Expected Values On-Drug Study
Status: Completed | Type: Observational
Sponsor: Accriva Diagnostics (Industry)
Responsible Party: Sponsor
Other Study IDs: VFN-CSS-16-0003
Record Dates: First submitted 2020-07-23; First posted 2020-07-30 (Actual); Last update posted 2020-07-30 (Actual); Status verified 2020-07

CONDITIONS: Coronary Disease; Platelet Aggregation
Keywords: aggregation; platelet; P2Y12 inhibitor; Aspirin
MeSH Terms: conditions — Coronary Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

GROUPS / COHORTS (2):
- Prasugrel: Patients taking prasugrel
  Interventions: Diagnostic Test: VerifyNow PRUTest
- Ticagrelor: Patients taking ticagrelor
  Interventions: Diagnostic Test: VerifyNow PRUTest

INTERVENTIONS:
Diagnostic Test: VerifyNow PRUTest — VerifyNow PRUTest for platelet aggregation

SUMMARY:
The purpose of this study is to determine the range of expected PRUTest values in patients in the intended use population receiving dual antiplatelet treatment with aspirin and prasugrel (Effient®), or ticagrelor (Brilinta®).

DETAILED DESCRIPTION:
The on-drug reference range study will be performed by measuring venous blood samples in duplicate collected from patients receiving prasugrel (Effient®), or ticagrelor (Brilinta®). Subjects must be on aspirin at the doses prescribed by their treating physician.

When possible, venous blood samples may be collected in conjunction with routine laboratory testing, to minimize the number of needle sticks for the subject. Alternatively, samples may be collected separately to complete the study.

A CBC measurement must be performed for each enrolled subject from a sample collected at the time of blood draw or within ± one week and tested at a certified laboratory. Samples for PRUTest collected in conjunction with a CBC must be drawn after the PRUTest sample.

Up to 130 subjects will be enrolled in the study to facilitate collection of the minimum number of blood samples needed to determine the on-drug reference range of prasugrel (Effient®), or ticagrelor (Brilinta®).

ELIGIBILITY:
Inclusion Criteria:

* • Males and females 18 years and older

  * Able and willing to provide written informed consent.
  * Current treatment with aspirin (any dose).
  * Have a planned or scheduled percutaneous coronary intervention (PCI) with the potential to receive treatment with prasugrel (Effient®), or ticagrelor (Brilinta®) following an oral loading dose or on maintenance treatment for a minimum of seven days who may have symptomatic cerebrovascular disease (transient ischemic attack or following a thrombotic stroke) or cardiovascular disease.

Exclusion Criteria:

* • Unable to provide written informed consent.

  * Currently receiving an investigational antiplatelet agent.
  * GP IIb/IIIa therapy (ReoPro®, Integrilin®, Aggrastat®) within the past 2 weeks.
  * Received any therapy containing dipyridamole (Persantine®, Aggrenox®) within the past 2 weeks.
  * Women who may be pregnant or are of child bearing potential

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Up to 130 subjects will be enrolled in the study to facilitate collection of the minimum number of blood samples needed to determine the on-drug reference range of prasugrel (Effient®), or ticagrelor (Brilinta®).
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2016-09-06 (Actual); Primary Completion 2017-08-14 (Actual); Study Completion 2018-03-22 (Actual)

PRIMARY OUTCOMES:
PRUTest | Within 24 hours of the loading or last maintance dose
  VerifyNow PRUTest results

CONTACTS AND LOCATIONS:
Overall Officials: Dominick J Angiolillo, M.D., Ph.D., Principal Investigator — Uunversity of Florida Health Jacksonville

IPD SHARING:
Plan to Share IPD: No
Publication of Results

REFERENCES:
- [Derived] Angiolillo DJ, Been L, Rubinstein M, Martin M, Rollini F, Franchi F. Use of the VerifyNow point of care assay to assess the pharmacodynamic effects of loading and maintenance dose regimens of prasugrel and ticagrelor. J Thromb Thrombolysis. 2021 Apr;51(3):741-747. doi: 10.1007/s11239-021-02386-7. Epub 2021 Feb 13. PMID 33582955